CLINICAL TRIAL: NCT02572921
Title: Evaluation of the Positive Psychotherapy to Reduce Symptoms and to Promote Happiness With Depressive Patients Compared to Cognitive-Behavioral Psychotherapy
Brief Title: Comparison of Positive Psychotherapy and Cognitive-Behavioral Psychotherapy for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Salzburg (Other)
Collaborators: The Wagner-Jauregg Provincial Neuropsychiatric Clinic (Individual)
Responsible Party: Principal Investigator, Mag. Linda Maria Furchtlehner, Principal Investigator, University of Salzburg
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: USalzburg
Record Dates: First submitted 2015-09-15; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Depression
Keywords: Positive Psychotherapy; Depression; Happiness
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive Psychotherapy (Experimental): Experimental Group (Positive Psychotherapy)
  Interventions: Behavioral: Positive Psychotherapy
- Cognitive Behavioral Therapy (Active Comparator): Active Control Group (Cognitive Behavioral Therapy)
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Positive Psychotherapy — The Positive Psychotherapy Group Treatment was developed by Martin Seligman and Tayyab Rashid (2013) and consists of 14 weekly group sessions of 2 hours. The strictly manualized program includes the following components:
  positive orientation and introduction, character strengths, signature strengths, good vs. bad memories, forgiveness, gratitude, satisficing vs. maximising, meaningful life, posttraumatic growth, hope and optimism, positive communication, signature strengths of others, savouring and slowness, altruism and the last session is about the integration of all these components to the "full life".
  Arms: Positive Psychotherapy
Behavioral: Cognitive behavioral therapy — This well-established, cognitive-behavior group therapy was developed by Schaub, Roth and Goldmann (2006) and consists of 12 weekly group sessions of 2 hours. The strictly manualized program includes the following components: education, building up activities, cognitive restructuring, relapse prevention. Moreover, there are 2 sessions added to the standard program: one session concerning savouring and the other one concerning stress reduction. Thus the whole program consists of 14 sessions.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study evaluates the effects of the Positive Psychotherapy on depressive symptoms and on happiness compared with regular cognitive behavioral therapy.

DETAILED DESCRIPTION:
Positive Psychotherapy (PPT) focuses on increasing well-being and positive emotions rather than ameliorating deficits in contrast to standard psychotherapy.

A lack of positive emotions, engagement and felt meaning are typically viewed as consequences or mere correlates of depression, while the PPT suggests that these may be causal for depression. Therefore building positive emotion, engagement and meaning will alleviate depression.

Thus PPT may offer a new way to treat and prevent depression.

The aim of this study is to compare the effects of the Positive Psychotherapy on depressive symptoms, life satisfaction and happiness in comparison to standard cognitive behavior psychotherapy (regular cognitive behavioral therapy).

60 mildly to moderately depressed patients are randomly assigned to the Positive Psychotherapy group or the regular cognitive behavioral therapy group.

Both treatments (primary intervention group and control group) are conducted in an outpatient group therapy setting with 14 sessions and a duration of 2-hours-per-week in small groups of 6 or 7 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Depression (Major depressive disorder, recurrent: mild to moderate; Major depressive disorder, single episode: mild to moderate; Dysthymic disorder)
* Patients should be between age 18 and 60

Exclusion Criteria:

* Any current treatment for depression
* Substance related or alcohol related disorder (within the last 12 months)
* Panic disorder
* Manic or hypomanic disorder
* Psychotic disorder * refusal to participate in a 14 weeks psychotherapy treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (measured by a self-report questionnaire) | fourteen weeks
  The depressive symptoms will be assessed by a self - report questionnaire: the Beck Depression Inventory II (BDI-II) which consists of 21 items
Depressive symptoms (measured by an assessment by others) | fourteen weeks
  The depressive symptoms will also be measured by an assessment by others: the Montgomery Asberg Depression Scale (MADS) which consists of 10 items
Happiness (measured by a self-report-questionnaire) | fourteen weeks
  Happiness will be assessed by a self-report-scale:
  the Flourishing-Scale (FS) which consists of 8 items
Happiness (measured by a self-report questionnaire) | fourteen weeks
  Happiness will be assessed by an additional self-report-questionnaire which consists of 25 items: the Positive Psychotherapy Inventory (PPTI)
Life satisfaction (measured by a self-report questionnaire) | fourteen weeks
  Life-Satisfaction will be measured by a self-report-questionnaire consisting of 5 items: the Satisfaction with Life Scale (SWLS)

SECONDARY OUTCOMES:
Clinical Symptoms | fourteen weeks
  Apart from depression also other clinical symptoms will be assessed by a self-report-scale with 53 items: the Brief Symptom Inventory (BSI)
Life events | six months
  Also life events will be assessed which happened during the last 6 months before starting the treatment and during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anton-Rupert Laireiter, Univ.-Prof.Dr., Study Chair — Paris Lodron University of Salzburg
Locations (2):
- Austria (2):
  - Beratungsstelle für Klinische Psychologie, Psychotherapie und Gesundheitspsychologie, Salzburg, Salzburg
  - Wagner-Jauregg- Hospital, Linz, Upper Austria